CLINICAL TRIAL: NCT03074604
Title: Carbon Dioxide Surgical Field Flooding and Aortic No-touch Off-pump Coronary Artery Bypass Grafting to Reduce Neurological Injuries After Surgical Coronary Revascularization (CANON): a Randomised, Controlled, Investigator and Patient Blinded Single Center Superiority Trial With Three Parallel Arms.
Acronym: CANON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Krzysztof Szwed, Dr., Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KB 60/2017
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Neurological Injury; Stroke; Postoperative Cognitive Dysfunction; Postoperative Delirium; Coronary Artery Disease; Coronary Artery Bypass Surgery; Off-Pump Coronary Artery Bypass
Keywords: Brain Injuries; Neurological Injury; Stroke; Postoperative Cognitive Dysfunction; Postoperative Delirium; Coronary Artery Disease; Coronary Artery Bypass Grafting; Coronary Artery Bypass Surgery; Bypass surgery; Beating Heart Coronary Artery Bypass; Off-Pump Coronary Artery Bypass
MeSH Terms: conditions — Trauma, Nervous System; Stroke; Postoperative Cognitive Complications; Emergence Delirium; Coronary Artery Disease; Brain Injuries

STUDY DESIGN:
Intervention Model Description: The CANON trial is designed as a randomised, controlled, investigator and patient blinded single center superiority trial with three parallel arms and a primary endpoint being the appearance of new lesions on control brain magnetic resonance imaging 3 days after surgery.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aortic no-touch OPCABG (Experimental): aortic no-touch OPCABG
  Interventions: Procedure: aortic no-touch OPCABG
- OPCABG with partial clamp applying carbon dioxide (Experimental): OPCABG with partial clamp applying carbon dioxide
  Interventions: Procedure: OPCABG with partial clamp applying carbon dioxide
- OPCABG with partial clamp (Active Comparator): OPCABG with partial clamp
  Interventions: Procedure: OPCABG with partial clamp

INTERVENTIONS:
Procedure: aortic no-touch OPCABG — (Study arm 1) In this intervention only the internal mammary artery grafts will be used (i.e. left internal mammary artery graft, right internal mammary artery graft, or a Y-graft that uses right internal mammary artery graft anastomosed onto left internal mammary artery graft to allow for a wide territory of myocardial revascularization). However, in the rare event that the aforementioned approach is insufficient to reach all target vessels, a reversed (great) saphenous vein graft may be used to extend the left internal mammary artery graft or the right internal mammary artery graft.
  Arms: aortic no-touch OPCABG
Procedure: OPCABG with partial clamp applying carbon dioxide — (Study arm 2) In this intervention chest cavity will be insufflated with carbon dioxide at a flow above 5 l/min during the entire surgical procedure.
  Arms: OPCABG with partial clamp applying carbon dioxide
Procedure: OPCABG with partial clamp — (Study arm 3) This is the control arm undergoing "traditional" OPCABG with partial clamp.
  Arms: OPCABG with partial clamp

SUMMARY:
The objective of this study is to investigate the value of employing the aortic no-touch off-pump coronary artery bypass technique and the practice of carbon dioxide surgical field flooding for the prevention of type 1 and 2 neurological injuries following surgical coronary revascularization.

DETAILED DESCRIPTION:
Neurological injuries remain a major concern following coronary artery bypass grafting (CABG) that offset survival benefit of CABG over percutaneous coronary interventions. Among numerous efforts to combat this issue, is off-pump CABG (OPCABG) that obviates the need for extracorporeal circulation and is associated with improved outcomes. The objective of this study is to examine whether the neuroprotective effect of OPCABG can be further pronounced by the use of two state-of-the-art operating techniques.

In this randomised, controlled, investigator and patient blinded single center superiority trial with three parallel arms a total of 360 patients will be recruited. They will be allocated in a 1:1:1 ratio to two treatment and one control arms. Treatment arms undergoing either aortic no-touch OPCABG or OPCABG with a partial clamp applying carbon dioxide surgical field flooding will be compared against control arm undergoing OPCABG. The primary endpoint will be the appearance of new lesions on control brain magnetic resonance imaging 3 days after surgery. Secondary endpoints will include the prevalence of new focal neurological deficits in the first 7 days after surgery, the occurrence of postoperative cognitive dysfunction at either 1 week or 3 months after surgery and the incidence of delirium in the first 7 days after surgery. Data will be analysed on intention-to-treat principles and a per protocol basis.

ELIGIBILITY:
Inclusion Criteria:

* elective and/or urgent coronary artery bypass

Exclusion Criteria:

* emergent and salvage setting
* score below age- and education-adjusted cut-off scores in mini mental state examination
* score above 8 on the subscales of hospital anxiety and depression scale
* neurologic deficit of any etiology
* previous psychiatric illness
* use of tranquilizers or antipsychotics
* alcohol or drug abuse
* history of cardiac surgery
* left ventricular ejection fraction less than 30%
* extracranial carotid artery stenosis of more than 70%
* body mass index of more than 35 kg/m2
* any contraindication for magnetic resonance imaging (e.g., magnetic resonance imaging - incompatible implantable device and claustrophobia)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
New lesions on control brain magnetic resonance imaging. | 3 days after surgery
  Appearance of new lesions on control brain magnetic resonance imaging 3 days after surgery.

SECONDARY OUTCOMES:
New focal neurological deficits. | 7 days after surgery
  Prevalence of new focal neurological deficits in the first 7 days after surgery.
Occurence of postoperative cognitive dysfunction | 1 week or 3 months after surgery
  Occurrence of postoperative cognitive dysfunction at either 1 week or 3 months after surgery
Incidence of delirium | 7 days after surgery
  Incidence of delirium in the first 7 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Szwed, M.D. Ph.D., Principal Investigator — Department of Clinical Neuropsychology, Nicolaus Copernicus University, Collegium Medicum, Poland; Alina Borkowska, Professor, Study Chair — Department of Clinical Neuropsychology, Nicolaus Copernicus University, Collegium Medicum, Poland
Locations (1):
- Department of Cardiac Surgery, Dr Antoni Jurasz Memorial University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, CSR
Time Frame: Available without time limits.
Access Criteria: The data that support the findings of this study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Krzysztof S, Wojciech P, Zbigniew S, Mariusz K, Remigiusz T, Damian P, Magdalena S, Marta T, Lech A, Alina B. CArbon dioxide surgical field flooding and aortic NO-touch off-pump coronary artery bypass grafting to reduce Neurological injuries after surgical coronary revascularisation (CANON): protocol for a randomised, controlled, investigator and patient blinded single-centre superiority trial with three parallel arms. BMJ Open. 2017 Jul 10;7(7):e016785. doi: 10.1136/bmjopen-2017-016785. PMID 28698347